CLINICAL TRIAL: NCT03595761
Title: Retrospective Study About 17 Cases of Child With Bacterial Meningitis Coupled With Cerebral Vasculitis
Brief Title: Meningitis With Cerebral Vasculitis in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0193
Record Dates: First submitted 2017-07-06; First posted 2018-07-23 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2017-07

CONDITIONS: Bacterial Meningitis
Keywords: cerebral vasculitis
MeSH Terms: conditions — Meningitis, Bacterial; Vasculitis, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purulent meningitis are life-threatening diseases in childhood. Cerebral vasculitis have been described in bacterial meningitis, but poor is known about their physiology and their impact on outcome.

The investigators decide to realize a retrospective mono-centric study carried out at Montpellier university hospital which looks back at a 7-year study(2009-2016).

The Investigators selected purulent meningitis cases based on the bacteriological data provided by the HDB (hospital data base). The Investigators divides in two groups : Group A if patients present a cerebral vasculitis ( radiologic diagnostic by RMI or tomodensitometry), in all, cases the diagnosis of vasculitis was confirmed by a radiologist specialised in neuropaediatrics by a second reading;Group B purulent meningitis with a cerebral vasculitis imaging.

Tuberculous meningitis, meningitis in CSF shunt, and in patients having chemotherapy were excluded.

The investigators report clinical and biological finding, inflammatory marker at the onset. The Investigators register also the clinical evolution and sequelae

DETAILED DESCRIPTION:
Meningitis steel are a cause of death in childhood. Cerebral complication are often responsable of poor prognosis. One of these complication vasculitis is steel not weel understood. There are only few study about it on children.

It is a retrospective study about 17 cases of chil which bacterial meningitis coupled wiethe cerebral vasculitis, the Investigators will describe epidemiology, bacteriology, evolution and corticosteroid treatment in this patients.

ELIGIBILITY:
Inclusion Criteria:

* bacterial meningitis with LCR confirmation

Exclusion criteria:

* tuberculous meningitis, immunosuppressor treatment, material like DVP

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with bacterial meningitis, and cerrbal vasculitis
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Found a difference demographic data | 1 day
  Found a difference demographic data between population A and B (age)
Found a difference demographic data | 1 day
  Found a difference demographic data between population A and B (gender)
Found a difference Clinical manifestation | 1 day
  Found a difference Clinical manifestation between population A and B
Found a difference Inflammatory parkers | 1 day
  Found a difference Inflammatory parkers between population A and B
Found a difference Infectious agent | 1 day
  Found a difference Infectious agent between population A and B

SECONDARY OUTCOMES:
Found a difference in the evolution of the diseases between group A and B | 1 day
  The data analysed will be : presence of seizure within the next 6 month before the last survey, necessity of antiepileptic treatment, development delay, presence of neurologic deficiency(palsy), persistence of abnormality on neuroimaging.
In the A group, studying the relationship between prescription of steroids pulse and final outcome and presence of sequelae. | 1 day
  Sequelae will be defined by the presence of one of this element : : presence of seizure within the next 6 month before the last survey, necessity of antiepileptic treatment, development delay, presence of neurologic deficiency(palsy), persistence of abnormality on neuroimaging.

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, Study Director — UH
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC